CLINICAL TRIAL: NCT05613348
Title: Humanized CAR19T2 T Cell in Children With Refractory/Relapsed B-cell Leukemia/Lymphoma
Brief Title: CD19 CAR T-cell Target Relapsed/Refractory Acute B Cell Leukemia/Lymphoma
Acronym: CAR19T2
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The company failed to provide corresponding CART services.
Sponsor: Zhujiang Hospital (Other)
Collaborators: Guangdong Zhaotai Cell Bio-tech Co., LTD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-KY-094
Record Dates: First submitted 2022-10-13; First posted 2022-11-14 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2022-10

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; B-Cell Lymphoma, Unspecified
Keywords: CAR T-cell; CAR19T2 T cell; refractory/relapsed B-cell acute lymphoblastic leukemia; refractory/relapsed Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, B-Cell; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- humanized CAR19T2 T cell to B-cell acute lymphoblastic leukemia/lymphoma (Experimental): Patients received fludarabine and cyclophosphamide (Flu/Cy) for lymphodepletion (Cy at 300-500 mg/m2/dose for four days and Flu at 20-30 mg/m2/dose for two days) before CAR19T2 T cells administration. This CAR19T2 T cell will be infused over 30 minutes on days Day 0.
  Interventions: Biological: CD19 CAR T-Cell(CAT19T2)

INTERVENTIONS:
Biological: CD19 CAR T-Cell(CAT19T2) — Drug: Fludarabine， Administered intravenously Drug: Cyclophosphamide， Administered intravenously

SUMMARY:
This study aims to evaluate the safety and efficacy of humanized Anti-CD19 Chimeric Antigen Receptor-T cell (CAR19T2 T cell) in children with refractory/relapsed B-cell acute lymphoblastic leukemia/lymphoma.

DETAILED DESCRIPTION:
CD19 CAR-T cells treating B-cell hematological malignancies have achieved unprecedented success. In this study, we investigated new third-generation autologous T cells (CAR19T2 T cells) genetically modified with humanized anti-CD19 construct incorporating CD28 and Toll-like receptor 2 (TLR2) costimulatory domains. CAR19T2 T cells will be modified before the infusion to those which could identify and kill the tumor cells (CD19+ cells). This study aims to evaluate the safety and efficacy of humanized Anti-CD19 Chimeric Antigen Receptor T cell (CAR19T2 T Cell) in children with refractory/relapsed B-cell acute lymphoblastic leukemia/lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. ≥1 year old and ≤18 years.
2. Patients with relapsed and/or refractory CD19-positive B-cell acute leukemia/lymphoma.
3. Leukemia/lymphoma relapsed after allogeneic hematopoietic stem cell transplantation within four weeks, all immunosuppressive agents were stopped for at least four weeks, and no active graft-versus-host disease(GVHD) was detonated.
4. Lansky play (≤16 years old) scale ≥60% or Karnofsky (>16 years old) score ≥60% and Eastern Cooperative Oncology Group (ECOG) performance status ≤1. Patients who are unable to walk because of paralysis, but who are up in a wheelchair will be considered ambulatory to assess the performance score.
5. Adequate vascular access leukapheresis procedure. Absolute Lymphocyte count (ALC) greater than or equal to 100 cells/μL.
6. Adequate renal, hepatic, pulmonary, and cardiac function is defined as the following:

   * Serum alanine aminotransferase/aspartate aminotransferase (ALT/AST) ≤ 5 upper limit of normal (ULN), Total bilirubin ≤2 x ULN.
   * A serum creatinine based on age/gender as follows: 1 to < 2 years: maximum serum creatinine 0.6 mg/dL (both male and female);2 to < 6 years: maximum serum creatinine 0.8 mg/dL (both male and female); 6 to < 10 years: maximum serum creatinine 1 mg/dL (both male and female); 10 to < 13 years: maximum serum creatinine 1.2 mg/dL (both male and female); 13 to < 16 years: maximum serum creatinine 1.5 mg/dL (male), 1.4 mg/dL (female); >=16 years: maximum serum creatinine 1.7 mg/dL (male), 1.4 mg/dL (female).
   * Baseline oxygen saturation > 92% on room air.
   * Echocardiogram or left ventricular ejection fraction (LVEF) greater than or equal to 45% confirmed by echocardiogram, no evidence of pericardial effusion (except trace or physiological), and no clinically significant arrhythmias.
7. Life expectancy of greater than or equal to 3 months.
8. Patients or legal guardians must sign an informed consent.

Exclusion Criteria:

1. Prior received any other CAR T cell and tumor vaccine treatment.
2. Patient with a previous history of active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection.
3. Patient with uncontrolled systemic fungal, bacterial, viral, or other infection (including tuberculosis) despite appropriate antibiotics or other treatment.
4. Acute GVHD grade II-IV (Glucksberg criteria) or chronic GVHD requiring systemic treatment within 4 weeks before enrollment.
5. History or presence of any CNS disorder such as a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, etc. (Except for CNS involvement of underlying hematological malignancy)
6. Severe psychological disorder or psychiatric illness.
7. Combined with life-threatening severe organ failure.
8. Major non-medicinal surgery within four weeks.
9. Received other clinical trials within four weeks. 10. Women who are pregnant or breastfeeding.

11. The following drugs patients must be stopped prior to leukapheresis:

* Tyrosine Kinase Inhibitor (TKI) must be discontinued more than or equal to 3 days before collection.
* Salvage chemotherapy must be stopped > 2 weeks and intrathecal chemotherapy in the 7 days prior to collection.
* Systemic steroid therapy exceeding the equivalent of 0.5 mg/kg/day of methylprednisolone in the 7 days before collection.
* Donor lymphocyte infusions (DLI) and Immunosuppressive therapies within 4 weeks before collection.
* Received clofarabine or cladribine within 3 months prior to collection.
* Receive blinatumomab within 4 weeks, inotuzumab ozogamicin, and rituximab within 4 months, and alemtuzumab within 6 months before collection.

  12. Tyrosine Kinase Inhibitor within 1 week and asparaginase within 4 weeks prior to CAR T-cell infusion.

  13. In the opinion of the PI, patients are present for any condition, not for enrollment.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 3 months
  A total number of patients achieved a Complete response (CR) or CR with incomplete blood count recovery (CRi) on Day 28 and three months by an independent review committee(IRC) assessment, as evaluated by peripheral blood, bone marrow, central nervous system (CNS) symptoms, physical exam (PE), and cerebrospinal fluid(CSF).
The maximum tolerated dose(MTD) of CAR19T2 T cells | 24 weeks
  The maximum tolerated dose(MTD) of CD19-positive relapsed/ refractory acute leukemia/lymphoma treated with CAR19T2 T cells.
Adverse Events (AEs) | 3 years
  Type, frequency and severity of adverse events (AEs), serious adverse events (SAE), and laboratory abnormalities (overall and in clinical, histological and molecular subgroups).

SECONDARY OUTCOMES:
Minimal residual disease (MRD) negative response rate | Up to 12 months after infusion
  Patients achieving CR or CRi and a negative MRD bone marrow.
Event-free survival (EFS) | Up to 3 years after infusion
  Time from CAR19T2 T cell infusion to progressive disease (PD), disease relapse, start of a new anticancer therapy, or death from any cause, whichever occurs first.
Overall survival (OS) | Up to 3 years after infusion
  Time from CAR19T2 T cell infusion to time of death due to any cause.
CAR-T cell expansion level | 24 months
  Copies numbers of CAR in peripheral blood (PB) and/or bone marrow (BM), CSF and lymph nodes, etc.
The duration of CAR T cell persistence | 24 months
  The duration of CAR T cell persistence in peripheral blood(PB) and/or bone marrow(BM), CSF and lymph nodes, etc.
Rate of hematopoietic stem cell transplant (HSCT) after CAR19T2 T cell infusion | Up to 3 years after CAR19T2 T infusion
  Percentage of subjects who achieve a response after CAR19T2 T cell infusion and then proceed to HSCT.
Maximum concentration of CAR19T2 T cell and cytokines. | 12 months
  Pharmacokinetics of CAR19T2 T cell in Maximum concentration.
Time to peak concentration of CAR19T2 T cell and cytokines. | 12 months
  Pharmacokinetics of CAR19T2 T cell in Time to peak concentration.
Area under the curve of CAR19T2 T cell and cytokines. | 12 months
  Pharmacokinetics of CAR19T2 T cell in Area under the curve.
Incidence of hypogammaglobulinaemia | 12 months
  Incidence and duration of hypogammaglobulinaemia.

CONTACTS AND LOCATIONS:
Overall Officials: Lihua Yang, Principal Investigator — Zhujiang Hospital
Locations (2):
- China (2):
  - Guangdong Zhaotai Cell Bio-tech Co., LTD, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guanzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No